CLINICAL TRIAL: NCT05816681
Title: An Open-label, Randomized, Multiple Dose, Parallel Study to Assess Elemental Impurities Level After Multiple Administration of DWJ1230 or DWB2001 in Subjects With Functional Diarrhea or Irritable Bowel Syndrome With Predominant Diarrhea(IBS-D)
Brief Title: Assessment of Elemental Impurities Level After Multiple Administration of DWJ1230 or DWB2001 in Subjects With Functional Diarrhea or Irritable Bowel Syndrome With Predominant Diarrhea.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DWJ1230101
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWJ1230 (Experimental)
  Interventions: Drug: DWJ1230
- DWB2001 (Experimental)
  Interventions: Drug: DWB2001

INTERVENTIONS:
Drug: DWJ1230 — Daewoong Pharmaceutical
  Arms: DWJ1230
Drug: DWB2001 — Daewoong Bio
  Arms: DWB2001

SUMMARY:
This study aims to assess elemental impurities level after dministration of dioctahedral smectite in subjects with functional diarrhea or irritable bowel syndrome with predominant diarrhea. Male or female subjects aged between 19 and 60 years will participate in the study. The study design is an opne-label, randomized, multiple dose paraller study. The patients were randomly assigned to DWJ1230 or DWB2001. It is intended that a total of 60 subjects will be enrolled to ensure that at least 24 subjects will complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic functional Diarrhea. (included Irritable Bowel Syndrome with perdominant diarrhea(IBS-D)).
* Male or Female subjects aged between 19 and 60 years at screening.
* Body Mass Index(BMI) between 18 and 27kg/m2 in male, 17 and 26kg/m2 in female. ※ BMI (kg/m2) = body weight (kg)/[height (m)]2
* Subjects who voluntarily decided to participate in the study and provided written consent to follow precautions after receiving a sufficient explanation on this study and fully understanding the information.

Exclusion Criteria:

* No history or clinically significant symptoms or severe disease, including cardiac, neurological, pulmonary, hepatic, biliary, gastrointestinal, endocrinologic, or renal disorders, or cancer.
* Identified or strongly suspected organic cause to diarrhea.
* Celiac disease or Intestinal malabsorption, Unspecified intestinal malabsorption.
* History of any serious adverse reaction or adverse event or hypersensitivity to any component of investigational product.
* Constipation, Iron deficiency anaemia, Hypocalcaemia, Osteoporosis.
* Known domestic, leisure or professional exposure to elemental impurities.
* Women who are breastfeeding or are planning to become pregnant during the study.
* Positive pregnancy test at screening.
* Presence of clinically significant physical, laboratory, vital signs, or ECG findings.
* Blood lead level > 3.3 μg/dL(=33.0 μg/L) at screening.
* galactose intolerance, fructose intolerance, Lapp lactase deficiency, sucurase-isomaltase deficiency, glucose-galactose malabsorption.
* Receipt of any investigational agent or study drug within 4 weeks prior to screening.
* Patients with history of alcohol or drug abuse.
* Subjects who donated whole blood within 2 months, donated blood components within 1 month.
* Subjects who have participated and taken investigational drug within 1 month prior to study drug administration.
* Subjects who the investigator considers inappropriate for the study due to other reasons.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
To assess the concentration of lead in blood after administration of Investigational Product | Day 7

SECONDARY OUTCOMES:
To assess blood concentration of other Class I(Cadmium, Arsenic, Mercury) after administration of Investigational Product | Day 7
To assess blood concentration of other Class IIa(Cobalt, Nickel) and of aluminium after administration of Investigational Product | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul ST. Mary's Hospital., Seoul, South Korea